CLINICAL TRIAL: NCT04294628
Title: Pilot Study of DS-8201a Pharmacodynamics in Patients With HER2-Expressing Advanced Solid Tumors
Brief Title: Testing the Biological Effects of DS-8201a on Patients With Advanced Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-01206; NCI-2020-01206 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-C-0154; P194688; 10346 (Other: National Cancer Institute LAO); 10346 (Other: CTEP)
Record Dates: First submitted 2020-03-03; First posted 2020-03-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Neoplasm; HER2-Positive Breast Carcinoma; Metastatic Malignant Solid Neoplasm; Refractory Malignant Solid Neoplasm; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (trastuzumab deruxtecan) (Experimental): Patients receive trastuzumab deruxtecan IV over 30-90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO or MUGA, CT or MRI, biopsies, and collection of blood samples throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Biological: Trastuzumab Deruxtecan

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Trastuzumab Deruxtecan — Given IV
  Other Names: DS-8201; DS-8201a; Enhertu; Fam-trastuzumab Deruxtecan-nxki; T-DXd; WHO 10516

SUMMARY:
This phase I trial studies the biological effects of DS-8201a on patients with HER2 positive cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). DS-8201a works by binding to a protein called HER2 that is present on the surface of tumor cells. This allows DS-8201a to kill the tumor cells by damaging their deoxyribonucleic acid (DNA), resulting in tumor cell death. This study looks at how DS-8201a may affect the levels of certain proteins and immune cells in tumors and how well the drug works against tumor cells by examining cells from a small piece tumor taken before and after DS-8201a is given.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the effects of trastuzumab deruxtecan (DS-8201a) on total Top1 levels in biopsy specimens from patients with HER2-expressing advanced solid tumors, at early and late post-treatment time points, thereby establishing the degree and duration of DS-8201 target engagement.

SECONDARY OBJECTIVES:

I. To assess any associations between serum concentrations of DS-8201a and the effects of DS-8201a on total Top1 levels in tumor biopsy specimens.

II. To determine the safety and tolerability of DS-8201a administered intravenously every 3 weeks, in 21-day cycles, at a dose of 5.4 mg/kg.

III. To determine the overall response rate (complete response [CR] + partial response [PR]) for patients administered intravenously with DS-8201a every 3 weeks, in 21-day cycles, at a dose of 5.4 mg/kg.

EXPLORATORY OBJECTIVES:

I. To evaluate the effects of DS-8201a on CD8+ T cell infiltration and activation in tumor, tumor PD-L1 and HER2 expression, and DDR signaling (for example: gamma H2AX, RAD51, and phosphorylated [p]NBS1) in biopsy specimens.

II. To examine genomic alterations in circulating tumor DNA (ctDNA) that may be associated with DS-8201a response or resistance.

III. To examine any associations between baseline tumor HER2 amplification or HER2 expression level and response to DS-8201a.

IV. To evaluate the effects of DS-8201a on tumor levels of HER2 and DDR-associated proteins.

V. To examine any tumor genomic alterations that may be associated with resistance to DS-8201a.

VI. To evaluate anti-drug antibodies following administration of DS-8201a.

OUTLINE:

Patients receive trastuzumab deruxtecan intravenously (IV) over 30-90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo echocardiography (ECHO) or multigated acquisition scan (MUGA), computed tomography (CT) or magnetic resonance imaging (MRI), biopsies, and collection of blood samples throughout the study.

After completion of study treatment, patients are followed up for 40 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Patients must have measurable or evaluable disease
* Age >= 18 years of age
* Patients must have HER2-positive or HER2-expressing tumors as defined by Clinical Laboratory Improvement Act (CLIA)-certified labs. Patients must have either:

  * A tumor HER2 immunohistochemistry (IHC) score of 1+ or greater (as determined by a CLIA-certified IHC test, per criteria specified) or
  * A tumor with HER2 amplification (as determined by CLIA-certified in situ hybridization [ISH] or a CLIA-certified next-generation sequencing assay)
* Patients with HER2 mutations are eligible, as are patients with HER2-positive breast cancer
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Absolute neutrophil count >= 1,500/mcL (within 8 days of enrollment)
* Platelets >= 100,000/mcL (within 8 days of enrollment)
* Leukocytes >= 3,000/mcL (within 8 days of enrollment)
* Hemoglobin >= 9 g/dL (>= 8.0 g/dL for gastric cancer [GC] only) (within 8 days of enrollment)
* Serum albumin >= 2.5 g/dL (GC only) (within 8 days of enrollment)
* Total bilirubin =< 1.5 x institutional upper limit of normal (=< 3 x upper limit of normal in the presence of documented Gilbert's syndrome or liver metastases at baseline) (within 8 days of enrollment)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal OR =< 5 x institutional upper limit of normal for patients with liver metastases at baseline (within 8 days of enrollment)
* Creatinine =< 1.5 x institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above 1.5 x institutional normal (within 8 days of enrollment)
* No transfusions with red blood cells or platelets are allowed within 1 week prior to screening assessment
* No administration of granulocyte colony-stimulating factor (G-CSF) is allowed within 1 week prior to screening assessment
* International normalized ratio (INR)/prothrombin time (PT) and either partial thromboplastin or activated partial thromboplastin time (aPTT) =< 1.5 x upper limit of normal (ULN)
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to provide blood samples for research purposes
* Patients must have a lesion or lesions amenable to biopsy and must be willing to undergo 3 core needle biopsy procedures for research purposes
* Patients must have left ventricular ejection fraction (LVEF) >= 50% by either an echocardiogram (ECHO), multigated acquisition (MUGA), or cardiac MRI scan within 28 days prior to enrollment
* Patients receiving standard of care androgen deprivation treatment (surgical castration versus luteinizing hormone-releasing hormone [LHRH] agonist or antagonist treatment) are eligible to participate in the trial. Patients receiving LHRH agonist or antagonist may continue treatment throughout the duration of this study
* Patients who are human immunodeficiency virus (HIV) positive may participate IF they meet the following eligibility requirements:

  * They must be stable on their anti-retroviral regimen, and they must be healthy from an HIV perspective
  * They must have a CD4 count of greater than 250 cells/mcL over the past 6 months on this same anti-retroviral regimen and must not have had a CD4 count < 200 cells/uL over the past 2 years, unless it was deemed related to the cancer and/or immunotherapy-induced bone marrow suppression

    * For patients who have received chemotherapy in the past 6 months, a CD4 count < 250 cells/ul during chemotherapy is permitted as long as viral loads were undetectable during this same chemotherapy
  * They must have an undetectable viral load and a CD4 count >= 250 cells/uL within 8 days of enrollment
  * They must not be currently receiving prophylactic therapy for an opportunistic infection and must not have had an opportunistic infection within the past 6 months HIV-infected patients should be monitored every 12 weeks for viral load and CD4 counts
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression for >= 1 month after treatment of the brain metastases
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* The effects of DS-8201a on the developing human fetus are unknown. For this reason and because HER2 antibodies conjugated to topoisomerase 1 inhibitor agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation and for at least 7 months after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of DS-8201a administration
* Women of non-child-bearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases, a blood sample with simultaneous follicle-stimulating hormone [FSH] > 40 mIU/mL and estradiol < 40 pg/mL [< 147 pmol/L] is confirmatory) are eligible. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods outlined for women of child-bearing potential if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method
* Subjects must not freeze, donate, or retrieve for their own use ova or sperm starting at screening, throughout the study period, and for at least 4.5 months after the final study drug administration. Preservation of sperm or ova should be considered prior to enrollment in this study
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with DS-8201a, breastfeeding should be discontinued if the mother is treated with DS-8201a

Exclusion Criteria:

* Patients who have had:

  * Chemotherapy (including antibody drug therapy, retinoid therapy, hormonal therapy for cancer-with the exception of standard of care androgen deprivation treatment) within:

    * 4 weeks or five half-lives, whichever is shorter, for small-molecule targeted agents such as 5-fluorouracil-based agents, folinate agents, weekly paclitaxel or
    * 6 weeks for nitrosoureas or mitomycin C or
  * Immunotherapy, including monoclonal antibody therapy, within 4 weeks
* Patients with any of the following pulmonary-related illnesses:

  * A history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, current ILD/pneumonitis, or for whom suspected ILD/pneumonitis cannot be ruled out by imaging at screening
  * Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (i.e., pulmonary emboli within three months of the study enrollment, severe asthma, severe chronic obstructive pulmonary disease [COPD] grade 3-4 per Global Initiative for Obstructive Lung Disease [GOLD] criteria, restrictive lung disease, pleural effusion, etc.), and any autoimmune, connective tissue, or inflammatory disorders with potential pulmonary involvement (i.e., Rheumatoid arthritis, Sjogren's, sarcoidosis, etc.), or prior pneumonectomy
* Patients who have had radiation therapy within 4 weeks (or palliative stereotactic radiation therapy within 2 weeks)
* Patients who have had a major surgery within 4 weeks
* Patients who are receiving any other investigational agents
* Patients with a medical history of myocardial infarction within 6 months before enrollment, symptomatic congestive heart failure (CHF) (New York Heart Association class II to IV), or with troponin levels consistent with myocardial infarction (as defined according to the assay manufacturer) 28 days prior to enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to DS-8201a (e.g., other topoisomerase I inhibitors) or the inactive ingredients in the drug product
* Patients who have a history of severe hypersensitivity reactions to other monoclonal antibodies
* Patients with a Fridericia's formula-corrected QT interval (QTcF) prolongation to > 470 ms (females) or > 450 ms (males) based on average of the screening triplicate 12-lead electrocardiogram (ECG)
* Patients with spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms
* Patients with an uncontrolled infection requiring IV antibiotics, antivirals, or antifungals
* Patients with unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to grade =< 1 or baseline. Subjects with chronic grade 2 toxicities (e.g., grade 2 chemotherapy-induced neuropathy) may be eligible per the discretion of the investigator after consultation with the sponsor medical monitor or designee. Subjects should no longer be symptomatic nor require treatment with corticosteroids or anticonvulsants and must have recovered from the acute toxic effect of radiotherapy
* Patients with substance abuse or any other medical conditions that would increase the safety risk to the subject or interfere with participation of the subject or evaluation of the clinical study in the opinion of the investigator
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because DS-8201a is a HER2 antibody conjugated to a topoisomerase 1 inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with DS-8201a, breastfeeding should be discontinued if the mother is treated with DS-8201a
* Patients are not allowed to receive chloroquine/hydroxychloroquine. Patients receiving chloroquine/hydroxychloroquine require a washout of > 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2027-01-19 (Estimated)

PRIMARY OUTCOMES:
Early topoisomerase 1 cleavable complex (Top1cc)/deoxyribonucleic acid (DNA) damage response (DDR) | Up to day 1 of cycle 3 (each cycle is 21 days) or optionally, up to time of disease progression or restaging follow-up
Tumor immune microenvironment response | Up to day 1 of cycle 3 (each cycle is 21 days) or optionally, up to time of disease progression or restaging follow-up

SECONDARY OUTCOMES:
Association between serum concentrations of DS-8201a and Top1cc formation | Up to day 1 of cycle 3 (each cycle is 21 days) or optionally, up to time of disease progression or restaging follow-up
  The association between serum concentrations of DS-8201a and Top1cc formation will be assessed by computing the sample correlation between the area under the DS-8201a serum concentration curve (AUC) and the initial change in Top1cc (from baseline to cycle 1 day 7 [C1D7]). Will also compute the sample correlation between the maximum serum concentration of DS-8201a and the initial change in Top1cc (from baseline to C1D7). These relationships will also be summarized graphically using scatterplots and overlaid LOWESS curves.
Incidence of adverse events | Up to 30 days post-treatment
  Descriptive analyses of Common Terminology Criteria for Adverse Events data will be performed, as will analysis of anti-drug antibodies.
Overall response rate | From the start of the treatment until disease progression/recurrence
  Will estimate the overall response rate (complete response + partial response) among eligible patients who have received at least one dose of DS-8201a. A 95% confidence interval for this response rate will also be computed. For this analysis, response classifications will follow Response Evaluation Criteria in Solid Tumors version 1.1 guidelines.

OTHER OUTCOMES:
Pharmacokinetic analysis | Cycle 1 day 1, prior to DS-8201a administration, at end of infusion, and at 5 hours post-infusion; at time of the cycle 1 day 7 biopsy; on day 1 of cycles 2, 3, and 4: prior to DS-8201a administration and at end of infusion
Pharmacodynamic analysis | Baseline, cycle 1 day 7, cycle 3 day 1, prior to DS-8201a administration, optionally at time of disease progression or "restaging follow-up"

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Shin, Principal Investigator — National Cancer Institute LAO
Locations (6):
- United States (6):
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - NYP/Weill Cornell Medical Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2024-11-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT04294628/ICF_000.pdf